CLINICAL TRIAL: NCT02697929
Title: Sugammadex Versus Neostigmine After Rocuronium Infusion During Liver Transplantation
Brief Title: Sugammadex/Neostigmine and Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Livia Pompei, MD, Azienda Ospedaliera S. Maria della Misericordia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SugNeoLTx1.0
Record Dates: First submitted 2016-02-13; First posted 2016-03-03 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Residual Curarization; Liver Transplantation
Keywords: Rocuronium
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugammadex (Active Comparator): at the end of surgery administration of 2 mg/kg of sugammadex after the third T2 twitch at Train of Four (TOF) stimulation
  Interventions: Drug: sugammadex
- neostigmine (Active Comparator): at the end of surgery administration of 50 mcg/kg of neostigmine after the third T2 twitch at Train of Four (TOF) stimulation
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: sugammadex
  Arms: sugammadex
Drug: Neostigmine
  Arms: neostigmine

SUMMARY:
Cirrhotic patients undergoing liver transplantation are at very high risk of post operative complication such as post-operative residual curarization.

Rocuronium is a neuromuscular blocking agent that nowadays can be safely and rapidly antagonized with sugammadex.

No one study compared sugammadex versus neostigmine after rocuronium infusion during liver transplantation.

DETAILED DESCRIPTION:
It is known that major abdominal surgery is associated with increased risk of morbidity and postoperative mortality. The complexity and the duration of the procedure as well as the failure to antagonize neuromuscular blocking agents at the end of surgical procedure are risk factors for postoperative complications.

Muscle relaxation plays an important role that is to facilitate intubation and to allow a better surgical condition. For this reason it is necessary to maintain, during the surgery, a deep neuromuscular block.

Deep block at the level of the adductor muscle of the thumb is obtained by measuring 1-2 responses during post-tetanic stimulation (the so-called Post-Tetanic Count or PTC).

The maintenance of a deep neuromuscular block requires further doses of neuromuscular blockers and, therefore, the need of long recovery times regardless of the drug used.

Pharmacodynamics and pharmacokinetics of neuromuscular blocking and reversals commonly used in clinical practice can undergo significant changes due to the presence of alterations in organ function such as hepatic and renal insufficiency. In these patients we see more frequent adverse events such as prolonged neuromuscular blockade and postoperative residual curarization.

In the literature it is considered suitable a recovery from neuromuscular block if the relationship between the fourth and first contraction during Train of Four (TOF) is greater than 0.9 (TOF-ratio> 0.9). This may take a long time so the reversal of blocking agents at the end of the surgical procedure is the solution to reduce this waiting period. The importance of an adequate recovery from neuromuscular block at the end of anesthesia is related to avoid postoperative residual paralysis (PORC) and reducing the risk of postoperative respiratory complications potentially fatal.

Rocuronium is characterized by an increase in half-life and an increase in the recovery time of neuromuscular transmission (TOF ratio of 0.9) in cirrhotic patients compared to controls healthy people.

To prevent residual neuromuscular blockade and all the complications that it brings with it it could be resorted the use of anti-cholinesterase drugs (neostigmine) to antagonize indirectly the action of non-depolarizing neuromuscular blocking agents. Neostigmine works by increasing the availability of acetylcholine at the neuromuscular junction. The administration of neostigmine may however cause bronchospasm, abdominal pain, nausea, cardiac arrhythmias and can not be used if the neuromuscular blockade is deep. Recently the use of sugammadex, a new drug that can act as an antidote to a comparison of non-depolarizing muscle relaxants amino-steroidal (rocuronium, vecuronium) showed good clinical impact. This drug works by encapsulating the muscle relaxant molecule in the plasma with a high affinity and binding to the complex thus formed which is then eliminated by the kidney. Sugammadex is characterized by the absence of adverse effects at the recommended doses and may be administered at correct dosage, even at deep neuromuscular blockade.

Several studies have shown that the recovery from neuromuscular blockade induced by rocuronium is significantly faster after administration of sugammadex compared with neostigmine both when used in moderate block levels and deep.

In literature there are no data and studies that assessed the recovery time of neuromuscular transmission (TOF ratio> 0.9) with the use of sugammadex verus neostigmine in patients undergoing liver transplantation after rocuronium infusion.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology status (ASA) III
* Ability to give a written informed consent
* Liver transplantation

Exclusion Criteria:

* Any allergy to medications involved in the study
* Any disease involving neuromuscular transmission
* Any therapy with toremifene, flucloxacillin or fusidic acid
* Renal disease with glomerular filtration rate less than 30 ml/min/1.73m2
* Hyperthermia maligna
* Anticonceptional therapy
* Pregnancy
* Core body temperature less than 35°C or skin temperature less than 32°C at the end of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Recovery time from moderate neuromuscular block to a TOF ratio more than 0.9 after administration of sugammadex or neostigmine using TOF-Watch SX. | 30 minutes

SECONDARY OUTCOMES:
Any episode PORC (defined as TOF ratio less than 0.9) within 20 minutes after extubation of the patient using TOF-Watch SX. | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: livia pompei, MD, Principal Investigator — AOU Santa Maria Della Misercordia; giorgio della rocca, FP, MD, Study Director — AOU Santa Maria Della Misercordia
Locations (1):
- AOU Santa Maria della Misericordia, Udine, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arbous MS, Meursing AE, van Kleef JW, de Lange JJ, Spoormans HH, Touw P, Werner FM, Grobbee DE. Impact of anesthesia management characteristics on severe morbidity and mortality. Anesthesiology. 2005 Feb;102(2):257-68; quiz 491-2. doi: 10.1097/00000542-200502000-00005. PMID 15681938
- [Background] Craig RG, Hunter JM. Neuromuscular blocking drugs and their antagonists in patients with organ disease. Anaesthesia. 2009 Mar;64 Suppl 1:55-65. doi: 10.1111/j.1365-2044.2008.05871.x. PMID 19222432
- [Background] van Miert MM, Eastwood NB, Boyd AH, Parker CJ, Hunter JM. The pharmacokinetics and pharmacodynamics of rocuronium in patients with hepatic cirrhosis. Br J Clin Pharmacol. 1997 Aug;44(2):139-44. doi: 10.1046/j.1365-2125.1997.00653.x. PMID 9278198
- [Background] Khalil M, D'Honneur G, Duvaldestin P, Slavov V, De Hys C, Gomeni R. Pharmacokinetics and pharmacodynamics of rocuronium in patients with cirrhosis. Anesthesiology. 1994 Jun;80(6):1241-7. doi: 10.1097/00000542-199406000-00011. PMID 8010470
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Derived] Deana C, Barbariol F, D'Inca S, Pompei L, Rocca GD. SUGAMMADEX versus neostigmine after ROCURONIUM continuous infusion in patients undergoing liver transplantation. BMC Anesthesiol. 2020 Mar 25;20(1):70. doi: 10.1186/s12871-020-00986-z. PMID 32213163